CLINICAL TRIAL: NCT00751738
Title: A Multi-center, Open-label, Follow-up Study to Assess the Long-term Safety of 125 mg Per Day of Oral Azimilide Dihydrochloride in Patients With an Implantable Cardioverter Defibrillator
Brief Title: Long Term Safety of 125 mg Per Day of Oral Azimilide in Patients With Implantable Cardioverter Defibrillator (ICDs)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Jose Brum, MD, Procter and Gamble Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001060
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — azimilide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 125 mg azimilide
  Interventions: Drug: azimilide dihydrochloride

INTERVENTIONS:
Drug: azimilide dihydrochloride — oral, once daily until sponsor stopped the study

SUMMARY:
This is an open-label, multi-center, long-term, (open-ended) safety study with 125 mg per day of azimilide in patients who completed protocol 2000098.

ELIGIBILITY:
Inclusion Criteria:

* patients who completed at least 12 months on study 2000098 before inclusion in this study

Exclusion Criteria:

* breast feeding or plan to become pregnant
* used ticlopidine
* were taking Class I or other Class III drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2002-10; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
safety of azimilide in this patient population | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Brum, MD, Study Director — Procter and Gamble
Locations (82):
- United States (46):
  - Research Facility, Mobile, Alabama
  - Research Facility, Little Rock, Arkansas
  - Research Facility, La Jolla, California
  - Research Facility, Loma Linda, California
  - Research Facility, Sacramento, California
  - Research Facility, Colorado Springs, Colorado
  - Research Facility, Bridgeport, Connecticut
  - Research Facility, Washington D.C., District of Columbia
  - Research Facility, Fort Lauderdale, Florida
  - Research Facility, Fort Myers, Florida
  - Research Facility, Jacksonville, Florida
  - Research Facility, Maywood, Illinois
  - Research Facility, Kansas City, Kansas
  - Research Facility, Portland, Maine
  - Research Facility, Baltimore, Maryland
  - Research Facility, Boston, Massachusetts
  - Research Facility, Burlington, Massachusetts
  - Research Facility, Worcester, Massachusetts
  - Research Facility, Warren Township, New Jersey
  - Research Facility, Brooklyn, New York
  - Research Facility, Johnson City, New York
  - Research Facility, New York, New York
  - Research Facility, Rochester, New York
  - Research Facility, West Orange, New York
  - Research Facility, Williamsville, New York
  - Research Site, Durham, North Carolina
  - Research Facility, Winston-Salem, North Carolina
  - Research Facility, Cincinnati, Ohio
  - Research Facility, Toledo, Ohio
  - Research Facility, Tulsa, Oklahoma
  - Research Facility, Erie, Pennsylvania
  - Research Facility, Hershey, Pennsylvania
  - Research Facility, Lancaster, Pennsylvania
  - Research Facility, Philadelphia, Pennsylvania
  - Research Facility, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Facility, Germantown, Tennessee
  - Research Facility, Nashville, Tennessee
  - Research Facility, Dallas, Texas
  - Research Facility, Houston, Texas
  - Research Facility, Salt Lake City, Utah
  - Research Facility, Charlottesville, Virginia
  - Research Facility, Fairfax, Virginia
  - Research Facility, Spokane, Washington
  - Research Facility, Green Bay, Wisconsin
  - Research Facility, Milwaukee, Wisconsin
- Belgium (2):
  - Research Facility, Bruges
  - Research Facility, Mont Godinne
- Canada (8):
  - Research Facility, Victoria, British Columbia
  - Research Facility, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Facility, Hamilton, Ontario
  - Research Facility, Ottawa, Ontario
  - Research Facility, Toronto, Ontario
  - Research Facility, Montreal, Quebec
  - Research Facility, Québec
- France (5):
  - Research Facility, Lille
  - Research Facility, Nantes
  - Research Facility, Paris
  - Research Facility, Pessac
  - Research Facility, Tours
- Germany (12):
  - Research Facility, Bad Bevensen
  - Research Facility, Berlin
  - Research Facility, Brandenburg
  - Research Facility, Coburg
  - Research Facility, Frankfurt
  - Research Facility, Freiburg im Breisgau
  - Research Facility, Hamburg
  - Research Facility, Heidelberg
  - Research Facility, Ludwigshafen
  - Research Facility, Magdeburg
  - Research Facility, Mannheim
  - Research Facility, Tübingen
- Poland (5):
  - Research Facility, Gdansk
  - Research Facility, Katowice
  - Research Facility, Lublin
  - Research Facility, Szczecin
  - Research Facility, Warsaw
- Spain (4):
  - Research Facility, Barcelona
  - Research Facility, Madrid
  - Research Facility, Málaga
  - Research Facility, Valencia